CLINICAL TRIAL: NCT06217614
Title: Beneficial Effects of Specific Natural Products on Management of Xerostomia: A Randomized Controlled Clinical Trial
Brief Title: Beneficial Effects of Natural Products on Management of Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-018
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Xerostomia; Diabetes Mellitus; Hypertension; Post COVID-19 Condition
Keywords: Manuka honey; Green tea; Natural products
MeSH Terms: conditions — Xerostomia; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Intervention Model Description: (Manuka honey-green tea) will topically be applied to the oral mucosa as oral rinse 3 times per day.
  Patients will be instructed not to swallow (Manuka honey-green tea) mouth rinse.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not know the intervention in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Manuka honey-green tea) interventional arm (Active Comparator): • (Manuka honey-green tea) will topically be applied to the oral mucosa as oral rinse 3 times per day to treat xerostomia.
  Interventions: Other: (Manuka honey-green tea)
- Saline mouthwash control group (Placebo Comparator): Patients in the control arm followed the same protocol with normal saline rinses in the same bottles 3 times per day for xerostomia
  Interventions: Other: (Manuka honey-green tea)

INTERVENTIONS:
Other: (Manuka honey-green tea) — Manuka honey is a natural honey, and green tea are herbs Dried green tea leaves (100 gm) will be soaked into 500 ml of methanol solution for two days. Green tea plus ginger mouthwash was prepared by adding 50% green tea extract and 50% ginger extract. After extraction, the extract was filtered and taker to the vacuum evaporator to remove the solvent.
  The mouthwash was prepared by adding 3 gm of each extract, 0.12 gm sodium saccharin, and one liter distilled water, then every 20 ml of Manuka honey were added in 100 ml of (green tea and ginger solution). Finally, the mixture was stirred vigorously until all the particles were dissolved. Thereafter the obtained mixture was filtered. The mouthwash then filled in sterilized amber color bottles of 250 ml each.
  According to similar studies performed in this field, the patients used a 20ml of (Manuka honey-green tea- ginger) mouthwash three times a day (preferably after their meals), kept it for one minute, and then poured it out

SUMMARY:
Xerostomia, the subjective feeling of oral dryness, is a symptom most frequently accompanied by either decreased salivary flow or an altered composition of saliva. Hyposalivation, on the other hand, is the objective measured reduction in salivary flow rate. Xerostomia is a relatively common complaint, particularly among older people, and can lead to major consequences with regard to the quality of their general and oral health and wellbeing.

Xerostomia has a variety of possible etiological factors; it is generally classified as having primary and secondary causes. Primary causes comprise conditions that directly affect the salivary glands and induce xerostomia like, Sjogren's syndrome, diabetes mellitus type 1 and 2, thyroid disease, adrenal pathology, renal or hepatic diseases, hepatitis C virus infection, and HIV disease.

DETAILED DESCRIPTION:
Multiple pharmacological and non-pharmacological measures that have been tested in previous studies in order to improve xerostomia in patients suffering from that complaint which were based on the stimulation of the salivary gland flow. Salivary glands can be stimulated to produce saliva mechanically (for example, by chewing gum, using different formulated mouthwashes or acupressure) or through medications (such as pilocarpine, cevimeline, angiotensin-converting enzyme inhibitors and angiotensin-receptor antagonists) Overall, the available interventions do not appear to provide an effective, comprehensive and long-term management of xerostomia. This has strengthened the need for further investigation of other interventions for the management of xerostomia As Egypt is considered a low-income country, therefore, the general properties of ideal saliva substitutes to be used should be inexpensive, edible, hydrating, safe-to-swallow but retainable in the mouth.

Given the importance of the oral health status of in patients suffering from dry mouth with the associated problems, and the limited availability of proper remedy for xerostomia in the Egyptian market. This study is designed to evaluate the efficiency of different and natural treatment as a mix of (Manuka honey -green tea) mouth rinse in management of xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* - Both genders, aged above 19 years.
* All patients must have complaint of xerostomia.
* Objective dry mouth score from (2-5).
* Subjective dry mouth score from (1-4).
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Patient with history of any serious illness as malignancy.
* Patients with any autoimmune disease.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in subjective dry mouth score | one month
  subjective dry mouth scores were calculated as the number of asked questions about dry mouth symptoms (0-4), and patients with a score higher than 1 considered having xerostomia so higher scores more than 1 out of 4 indicating xerostomia but lower scores suggesting improvement.

SECONDARY OUTCOMES:
Changes in objective dry mouth score | one month
  Objective dry mouth scores were calculated as the number of observed dry mouth signs (0-5), and patients with a score higher than 2 having xerostomia so higher scores more than 2 out of 5 indicating xerostomia but lower scores suggesting improvement
Salivary flow rates | one month
  Eating and talking were prohibited during the time of collection. Unstimulated whole saliva was collected for 5 min by spitting method. The collection will be timed, so that flow rate (mL/min) could be measure.
  increasing in the salivary flow rate of the unstimulated saliva is considered improvment
Salivary Nitric oxide levels | one month
  Increasing in the salivary nitric oxide levels indicating improvment

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Egypt